CLINICAL TRIAL: NCT06804967
Title: Effects of Virtual Reality Relaxation on the Anxiety Levels of Adolescents and Adults During Orthodontic Bonding: A Randomized Controlled Trial
Brief Title: Effects of Virtual Reality Relaxation on the Anxiety Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Hakan Turkkahraman, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25009
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anxiety
Keywords: dental anxiety; orthodontic anxiety; virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Virtual Reality Relaxation Headset (Experimental): The experimental group will use Virtual Reality Relaxation (VRR) during the procedure. Meta Quest 3 is a virtual reality headset featuring an adjustable, pre-installed Standard Facial Interface. It comes with two Touch Plus Controllers with wrist straps. However, to prevent gamification and interaction, hand controllers will not be provided to participants to maintain uniformity in the virtual reality experience. Participants will be restricted from engaging in active movement or interacting with the software. The headset is lightweight, weighing just over one pound, and includes a soft, adjustable strap designed to fit various head shapes and hairstyles for added comfort. It also features built-in stereo speakers with 3D spatial audio for an immersive experience. Patients will receive brief instruction on how to comfortably position and adjust the headset as well as adjust the volume.
  Interventions: Device: virtual reality relaxation headset
- No intervention (No Intervention): Subjects in this group will not use the headset or any other form of intervention

INTERVENTIONS:
Device: virtual reality relaxation headset — No headset will be used
  Other Names: no intervention
  Arms: Virtual Reality Relaxation Headset

SUMMARY:
The goal of this clinical trial is to determine the effects of virtual reality relaxation on dental anxiety levels of adolescents and adults during an orthodontic bonding procedure.

The specific aim is to compare changes in the anxiety levels based on 1) psychological outcomes and 2) physiological outcomes between patients who experienced (virtual reality relaxation) VRR intervention during the orthodontic bonding procedure and those in the control group who did not receive the intervention

After provding written consent, subjects will be randomized to either the virtual reality device usage during their bonding procedure or no virtual reality device. They will have vital signs taken/anxiety level measured and answer a questionnaire before and after the device/no device usage (30 minutes).

DETAILED DESCRIPTION:
On the day of the bonding procedure, informed consent will be obtained from participants and parents/guardians who were not present during the treatment plan presentation appointment. Pre-operative data will be collected, prior to the start of orthodontic treatment. Once the patient is seated, a timer will be set for 5 minutes to allow the patient to recover and get settled in before measurements are taken. After this 5-minute period, the following measurements will be collected: (1) Vitals will be recorded with the patient seated in the upright position, including maximal blood pressure (BP) using Omron 3 series upper arm blood pressure monitor with cuff on the participant's right bicep, and heart rate (HR) and oxygen saturation (SpO2) using Masimo MightySat fingertip pulse oximeter on the right ring finger; (2) The patient's state anxiety will be evaluated through the completion of the five-item state form of Spielberger's State-Trait Anxiety Inventory (STAIS-5); and (3) The patient's current anxiety level will be assessed by completing the Visual Analog Scale for anxiety (VAS-A).

The provider will review with the experimental group participants the purpose of VR and explain in a calm and soothing tone that using VR during dental procedures has been found to relax patients and to reduce their blood pressure and heart rate while also at times increasing oxygen levels. For patients in the experimental group, they will be told they will be immersed in VR for a maximum of 30 minutes. During this time period, one arch, either maxillary or mandibular, will be bonded.

Following the general explanation about the use of VR within a dental procedure, a written list with corresponding visual representation of the available virtual environments (VE) from Nature Treks will be provided (e.g. Orange Sunset, White Winter, Red Savanna). Patients will be requested to choose their preferred VE to experience during the procedure. The investigator will launch the Nature Treks application, hand the headset to the patient to put on, and assist them in adjusting the straps for a comfortable fit. A brief window of approximately 30-60 seconds will be given for them to acclimate to the virtual surroundings and to also confirm the patient's desire to proceed. During this short period, patients will be offered the choice to alter the setting or remain in it for the designated 30-minute duration. The environment selected by patients will be recorded and stored in RedCap. Participants in the control group will not be provided with the VR headset during the procedure and will have full visibility of the clinic area.

Once all relevant questions are answered, the patient will be reclined in the dental chair. The 30-minute timer will start when the orthodontic resident initiates the orthodontic bonding procedure by placing the cheek retractor for isolation.

Post-operative data will be collected 30 minutes after the start of the procedure for both groups. At the 30-minute mark, the procedure will be paused, regardless of whether the entire arch has been bonded, and all correctly positioned brackets will be light-cured to allow for the removal of isolation. The patient will then be positioned upright, and the VR headset will be removed from the experimental group. T1 data will be collected immediately, including the (1) BP, HR, and SpO2, (2) the STAIS-5 completed form, and (3) the VAS-A completed form.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for fixed orthodontic treatment at IUSD Graduate Orthodontic Clinic
* Comprehensive treatment case
* Maxillary or mandibular arch bonding
* Patients > 13 years of age
* Must be able to read written English and comprehend spoken English

Exclusion Criteria:

* Re-treatment cases
* Diagnosed and/or reported clinical general anxiety disorder
* Currently taking pharmacologic anxiolytics
* Light hypersensitivity
* Self-reported history of seizures, concussions
* History of moderate to severe clinically diagnosed mental illness
* Self-reported history of hypertension or severe heart disease
* Self-reported history of a cardiac pacemaker or defibrillator
* Visual and/or auditory impairment
* Patients with craniofacial anomalies
* History of significant motion sickness or vertigo

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory (STAI-6) | Baseline (Before bonding procedure) and 30 minutes.
  State anxiety targets how a person feels at a specific moment while trait anxiety examines how a person usually feels. Both forms consist of anxiety-present items such as "I feel secure", and anxiety absent items, such as "I feel tense." Lower scores indicate for the purposes of this study, we will only administer the state anxiety questionnaire to determine the change in patients' anxiety levels in the dental setting.
Visual analog scale for anxiety (VAS-A) | Baseline (Before bonding procedure) and 30 minutes.
  The scale consists of a horizontal line with 'no anxiety' indicated on the left and 'worst possible anxiety' on the right. Subjects will be asked to mark (X) on the scale that best describes how they are feeling at the current moment. 0 represents not anxious at all and 10 represents extremely anxious.

SECONDARY OUTCOMES:
Blood pressure (BP) | Baseline (Before bonding procedure) and 30 minutes.
  Blood pressure (BP) of the subjects will be measured and collected using a Omron 3 series upper arm blood pressure monitor. This physiological metric will serve as a secondary outcome measure of anxiety and will be used to provide comparative data alongside the self-reported assessments.
Heart Rate (HR) | Baseline (Before bonding procedure) and 30 minutes.
  Heart Rate (HR) of the subjects will be measured and collected using a Omron 3 series upper arm blood pressure monitor. This physiological metric will serve as a secondary outcome measure of anxiety and will be used to provide comparative data alongside the self-reported assessments.
Oxygen Saturation Level (SpO2) | Baseline (Before bonding procedure) and 30 minutes.
  Oxygen Saturation Level (SpO2) of the subjects will be measured and collected using a a Masimo MightySat fingertip pulse oximeter. This physiological metric will serve as a secondary outcome measure of anxiety and will be used to provide comparative data alongside the self-reported assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Turkkahraman, DDS, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry Department of Orthodontics and Oral Facial Genetics Grad Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the HIPAA regulations.